CLINICAL TRIAL: NCT05376046
Title: Study of Erythrocyte Parameters and Hypercoagulability in Sickle Cell Disease
Brief Title: Study of Erythrocyte Parameters and Hypercoagulability in Sickle Cell Disease (SCD-TGA)
Acronym: SCD-TGA
Status: Recruiting | Type: Observational
Sponsor: BILLOIR (Other)
Responsible Party: Sponsor-Investigator, BILLOIR, Associate Professor, University Hospital, Rouen
Organization: University Hospital, Rouen (Other)
Other Study IDs: 2021/0328/OB
Record Dates: First submitted 2022-04-29; First posted 2022-05-17 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis
Keywords: sickle cell disease; vaso-occlusive crisis; reticulocyte count; thrombin generation assay; hypercoagulability
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sickle cell disease: Confirmed sickle cell disease withHaemoglobin profile was determined by high performance liquid chromatography (HPLC) (Variant II Biorad, California, United States), by capillary electrophoresis on Capillarys 3 Octa® (Kit hydragel hémoglobine Sebia, Lisses, France) and iso-electrofocalisation.
  Patients were included during injury evaluation in our tertiary centre.
  Interventions: Biological: Erythrocytic parameters and thrombin generation assay measurement
- Healthy: 25 healthy controls matched on age and gender
  Interventions: Biological: Erythrocytic parameters and thrombin generation assay measurement

INTERVENTIONS:
Biological: Erythrocytic parameters and thrombin generation assay measurement — Erythrocytic parameters and thrombin generation assay measurement

SUMMARY:
Sickle cell disease (SCD) is an inherited haemoglobinopathy disorder caused by mutations in HBB gene with amino-acid substitution on β globin chain. The consequence is synthesis of altered haemoglobin S (HbS) which polymerises in red blood cell (RBC) at deoxygenated state. SCD is associated with chronic haemolytic anaemia, vaso-occlusive crisis (VOC) leading to frequent hospitalisation.

The aim of the study was to to investigate whether a combination of routine laboratory biomarkers of haemolysis could be used to predict VOC development in confirmed SCD patients.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease

Exclusion Criteria:

* <18 years
* pregnancy
* Patient under protective guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients in the study were diagnosed and treated for SCD at Rouen University Hospital. Patients were included during annual visit in our tertiary centre. Patients with VOC were included less than 24hours after admission to emergency department. All patients treated with hydroxyurea have been treated for at least three years. All patients received a systematic annual visit to determine VOC development in the year. Patients were analyzed in four subgroups based on genotype and clinical status:
  * homozygous SCD (S/S) or β0 thalassemia (S/β0) at steady state;
  * homozygous SCD with α3.7 thalassemia (S/Sα3.7) at steady state;
  * heterozygous SCD with C haemoglobin (S/C) or β+ thalassemia (S/β+)at steady state;
  * patients hospitalized for VOC with any genotype.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalisation for Vaso-occlusive crisis within one years | 1 year
  Following injury consultation, evaluation of biological markers predicting vaso-occlusive crisis requiring hospitalisation in the year

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen university Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feugray G, Grall M, Gillardin B, Burdeau J, Ozanne N, Dumesnil C, Fauvel C, Billoir P. Hemoglobin and High-Density Lipoprotein as Biomarker of Left Atrial Dilatation in Sickle Cell Disease. EJHaem. 2025 Aug 22;6(4):e70135. doi: 10.1002/jha2.70135. eCollection 2025 Aug. PMID 40862241